CLINICAL TRIAL: NCT03991039
Title: Treatment of Primary Trigeminal Neuralgia: A Comparative Study of Microvascular Decompression and Stereotactic Gamma Knife Radiosurgery
Brief Title: Comparing Clinical Benefits of Gamma Knife and Microvascular Decompression for Trigeminal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Dr. Moneer k. Faraj, Consultant neurosurgeon, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neurosciences-iraq
Record Dates: First submitted 2019-06-15; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Trigeminal Neuralgia
Keywords: Trigeminal neuralgia, treatment
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Radiosurgery; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamma knife group (Active Comparator): Patients selected to be treated with gamma knife radiosurgery
  Interventions: Radiation: Gamma knife
- MVD Group (Active Comparator): Patients treated with microvascular decompression
  Interventions: Radiation: Gamma knife

INTERVENTIONS:
Radiation: Gamma knife — Microvascular decompression
  Other Names: Surgery

SUMMARY:
Clinical randomized study to compare the clinical effectiveness between two modalities of treatment of trigeminal neuralgia namely gamma knife radio surgery and microvascular decompression

DETAILED DESCRIPTION:
A randomized prospective study conducted in The Neurosciences Hospital, Baghdad, from January 2016 to January 2018, patients had either GKR treatment or treated with MVD. The pain evaluated pre- and post-operatively using the Barrow Neurological Institute Pain Intensity scale (BNIPI), visual analog scale (VAS) and Brief Pain Inventory Facial (BPI-Facial) scoring systems. In GKR procedure, the trigeminal root entry zone targeted with a radiation dose of 80 Gy. MVD was performed using retro-sigmoid approach. Follow-up period for two years

ELIGIBILITY:
Inclusion Criteria:

* primary idiopathic trigeminal neuralgia

Exclusion Criteria:

* secondary trigeminal neuralgia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Barrow Neurological Institute Pain Intensity scale (1-5) | Two years
  The pain evaluated pre- and post-operatively with the use of analgesic drugs the best is 1 indicates free of pain, the worst is 5. It is dependent score
visual analog scale (0-10) | Two years
  Pain severity described subjectively by the patient himself pre and post treatment , the 0 is free of pain and worst is 10. It is dependent score
Brief Pain Inventory (1-7) | ُTwo years
  Assess pain severity as impact to functional activities, the 7 is normal live activity and the worst is 1. It is dependent score

CONTACTS AND LOCATIONS:
Overall Officials: Moneer K. Faraj, Facs, Principal Investigator — Neurosciences hospital

IPD SHARING:
Plan to Share IPD: No